CLINICAL TRIAL: NCT05131516
Title: Ability of Peripheral Venous Pressure Variation to Predict Fluid Responsiveness During an Alveolar Recruitment Maneuver in Patients Undergoing Non Cardiac Surgery
Brief Title: Peripheral Venous Pressure Variation and Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Université Paris-Saclay-Assistance publique des hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Study PI, Erasme University Hospital
Other Study IDs: IRBN902021/CHUSTE
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Fluid Responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Alveolar recrutment maneuver — alveolar recruitment maneuver (30 mmHg for 30 seconds)

SUMMARY:
The decision to give fluids or not should not be taken lightly. Indeed, excessive or insufficient fluid administration is associated with increased morbidity and mortality. Prediction of fluid responsiveness relies on the use of a hemodynamic variable to determine how likely a patient is going to respond to a fluid bolus with a significant increase in their cardiac output or stroke volume. Depending on the response to fluids, patients are either responders or non-responders.

Today, we have many techniques to predict fluid responsiveness. However, almost all require the use of an advanced hemodynamic monitoring device.

DETAILED DESCRIPTION:
Predicting fluid responsiveness is important in the operating room in order to avoid unnecessary fluid administration. Over the last 15 years, a number of dynamic tests have been developed which are based on the principle of inducing short-term changes in cardiac preload, using heart-lung interactions, the passive leg raise or by the infusion of small volumes of fluid, and to observe the resulting effect on cardiac output or stroke volume. Pulse pressure and stroke volume variations were first developed, but they are reliable only under strict conditions. The variations in vena caval diameters share many limitations of pulse pressure variations. The passive leg-raising test is now supported by solid evidence and is more frequently used but not practical in the operating room. More recently, the end-expiratory occlusion test has also been described, which is easily performed in ventilated patients. Unlike the traditional fluid challenge, these dynamic tests do not lead to fluid overload. The dynamic tests require the insertion of an arterial catheter linked to an advanced cardiac output monitoring device which is costly and not applicable in lower risk patients without an arterial line.

In the operating room, it is recommended to use alveolar recruitment maneuvers, consisting in the transient administration of higher pressure levels, allowing to re-ventilate certain pulmonary territories by re-expanding alveoli that would have collapsed under mechanical ventilation. In daily practice, it is generally accepted that a patient presenting a significant fall in stroke volume or mean arterial pressure during an alveolar recruitment maneuver is preload dependent, but the scientific evidence in the literature remains insufficient to date. A previous study has also demonstrated the ability to predict fluid responsiveness via analysis of central venous pressure during a recruitment maneuver. By extrapolation, we would like to evaluate the capacity of peripheral venous pressure to predict this fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients scheduled for a high-risk abdominal surgery
* Patients equipped with an arterial line connected to an cardiac output hemodynamic monitoring device ( Flotrac, EV1000, Edwards Lifesciences, Irvine, USA)
* Patients in whom a recrutment maneuver is planned as per standard of care

Exclusion Criteria:

* Arythmia ( atrial fibrillation)
* Right ventricular dysfunction

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a high-risk abdominal surgery ( liver resection and pancreatectomy)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Ability of the peripheral venous pressure to predict fluid responsiveness | during surgery
  we will induce, before skin incision, an alveolar recrutment maneuver (standard of care) and observe variations of peripheral venous pressure, then, it will be followed by a volume expansion of 4ml/kg over 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDRE JOOSTEN, MD PhD, Principal Investigator — ERASME
Locations (1):
- ALEXANDRE joosten, Villejuif, France

IPD SHARING:
Plan to Share IPD: No